CLINICAL TRIAL: NCT02766907
Title: Optimizing the Ocular Surface Prior to Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioTissue Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P015-2
Record Dates: First submitted 2016-04-25; First posted 2016-05-10 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Corneal Dystrophy, Epithelial Basement Membrane
MeSH Terms: conditions — Corneal dystrophy, epithelial basement membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study (Active Comparator): prospective arm receiving cryopreserved amniotic membrane
  Interventions: Device: cryopreserved amniotic membrane
- Control (No Intervention): Retrospective review of debridement without cryopreserved amniotic membrane

INTERVENTIONS:
Device: cryopreserved amniotic membrane — placement of cryopreserved amniotic membrane after routine debridement procedure for EBMD
  Other Names: Prokera Slim (PKS)
  Arms: Study

SUMMARY:
Prospective study to evaluate the efficacy of using self-retained cryopreserved amniotic membrane after debridement in treating Epithelial Base Membrane Dystrophy (EBMD) to optimize the ocular surface integrity and intraocular lens calculation before cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with significant EBMD that are contemplating cataract surgery.
2. Age range: 50 years and older.
3. Both Genders and all ethnic groups comparable with the local community.
4. Subjects able to understand and willing to sign a written informed consent.
5. Subjects able and willing to cooperate with the investigational plan.
6. Subjects able and willing to complete postoperative follow-up.

Exclusion Criteria:

1. Subjects with known intolerance to PKS or known allergy to its preservative media.
2. Subjects with symblepharon or lid abnormality preventing PKS placement.
3. Ocular infection within 14 days prior to study entry.
4. Previous ocular surgery or injury within 3 months before enrollment.
5. Subjects with a history of non-healing epithelial defect or neurotrophic keratitis.
6. Inability or unwillingness of subject to give written informed consent, follow investigational plan or complete postoperative follow-up.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2017-01 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Yeu, MD, Principal Investigator — Virginia Eye Consultants
Locations (1):
- Virginia Eye Consultants, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study: prospective arm receiving cryopreserved amniotic membrane
  cryopreserved amniotic membrane: placement of cryopreserved amniotic membrane after routine debridement procedure for epithelial basement membrane dystrophy (EBMD)
Period: Overall Study
Arm/Group | Control | Study
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study | Control | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (7.5) | 66.5 (5.9) | 70 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Lens Calculation
Description: Assessed by corneal topography
Time Frame: Change from Baseline to 1 month
Measure: Mean (Standard Deviation); unit: D
Arm/Group | Study | Control
Number analyzed (Participants) | 9 | 9
D | 1.56 (1.6) | 0.94 (0.7)

2. Primary Outcome: Change in Intraocular Lens Power Calculation
Description: Assessed using biometry and calculated using Holladay I formula
Time Frame: Change from Baseline to 1 month
Measure: Mean (Standard Deviation); unit: D
Arm/Group | Study | Control
Number analyzed (Participants) | 9 | 9
D | 1.18 (1.2) | 0.79 (0.5)

ADVERSE EVENTS:
Arm/Group | Study | Control
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No